CLINICAL TRIAL: NCT06334029
Title: Observational Study of the Structural-functional Connectome in Patients With Epilepsy
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 12.2022
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Epilepsy: Recording of resting state EEG and MRI
  Interventions: Diagnostic Test: Functional and structural Connectome
- Control group: EEG resting state data recording
  Interventions: Diagnostic Test: Functional and structural Connectome

INTERVENTIONS:
Diagnostic Test: Functional and structural Connectome — Reconstruction of EEG derived functional relationship between brain regions (functional connectome). Reconstruction of thickness covariance across brain regions (structural connectome)

SUMMARY:
Over the past decade, the concept of the brain as a complex network has extremely influenced the way regarding how the latter is studied (Bartolomei et al., 2017). The structure of both structural and functional networks within the brain has been related to optimal brain functioning (Duma et al., 2022). This evolution of methods and approaches of investigation has directly impacted the study of epilepsy. An early conception of focal epilepsy was that it was related to the activity of the epileptogenic zone, which was identified as the generative element of seizures. However, what was previously considered focal was found to be network alterations at various levels, thus moving from the epileptogenic zone to the concept of the epileptogenic network. Alterations in both the structural and functional network, compared with a healthy control population, have been identified in various forms of epilepsy from focal to idiopathic generalized epilepsy (Lariviere et al., 2022, Zhang et al., 2009). Often the identification and removal of the epileptogenic network, turns out to be the elective therapy in drug-resistant focal epilepsies. The process of diagnosing and defining the epileptogenic network is still debated today. One of the most widely used methods is the implantation of intracranial electrodes for electroencephalographic recording of seizures (Bartolomei et al., 2017). This methodology carries with it several, albeit controlled, risks to the patient. New noninvasive approaches are being developed seeking to integrate information from structural neuroimaging and cortical electrical activity measured by high-density electroencephalography with external electrodes (Duma et al., 2021). These new approaches also include simulative approaches that exploit individualized information such as cortex geometry and patient-specific white matter connections (Courtiol et al. 2020). Thus, starting from a simple structural and diffusion MRI, which is done in routine clinical examinations, multiple localizing hypotheses of the epileptogenic network can be tested using simulative models and then compared with the real EEG signal as validation. Of great relevance is also to understand how the structural-functional connectome relates to cognitive function in patients with epilepsy, who have a high probability of presenting impaired functioning in one or more cognitive domains.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of focal or generalized epilepsy confirmed by specialist evaluation;
* at least one MRI scan of the brain that includes T1w
* at least one recording with resting state EEG
* age between 6 and 65 years at the time of the evaluation of the present study;
* ability to take part in a neuropsychological assessment.

Exclusion Criteria:

* vascular causes or non-low grade tumors as causes of epilepsy
* age different from the range 6-65 years
* neuroradiologic examination not complete
* absence of resting state recording
* inability to take part in a neuropsychological evaluation.

Ages: 6 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with focal epilepsy with drug resistance
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2026-11-22 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of regional alteration in the value of functional connectivity | once at recrutiment
  By comparing the value of functional connectivity derived from the EEG, between Epilepsy and control group, it is possible to identify altered brain regions to non-invasively identify the epileptogenic area, improving the diagnostic process

SECONDARY OUTCOMES:
Measuring the spread of the epileptogenic network | once at recrutiment
  In the Epilepsy group the correlation between the functional and the structural connectome identify the spreading of the epileptogenic network, and therefore the intensity of the pathology, guiding the diagnostic process

OTHER OUTCOMES:
Correlation between the Rey Complex figure test and the regional functional alteration | once at recrutiment
  The correlation between the Rey complex figure test measuring the memory efficiency and the regional functional connectivity provides a potential diagnostic tool helping the identification of the alteration of brain areas in relationship to the known impairment of memory in patients with epilepsy

CONTACTS AND LOCATIONS:
Overall Officials: Gian Marco Duma, PhD, Principal Investigator — IRCCS E. Medea
Locations (1):
- IRCCS E.Medea, Conegliano, Treviso, Italy

IPD SHARING:
Plan to Share IPD: No